CLINICAL TRIAL: NCT05077540
Title: The Effect of Oxytocin Versus, Sublingual Misoprostol in the Secondary Prevention of Postpartum Hemorrhage After Vaginal Delivery: a Randomized Controlled Trial
Brief Title: Oxytocin Versus, Sublingual Misoprostol in the Secondary Prevention of Postpartum Hemorrhage After Vaginal Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Clinical Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/543/8/21
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Labor Complication
MeSH Terms: conditions — Obstetric Labor Complications | interventions — Oxytocin; Misoprostol

STUDY DESIGN:
Intervention Model Description: double-blinded a randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded a randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxytocin (Active Comparator): 20 unit of oxytocin infusion in 500 ml lactated ringer's solution 125 ml/h (Syntocinon, Novartis, Switzerland)
  Interventions: Drug: oxytocin
- misoprostol (Experimental): 800 µg sublingual misoprostol (Cytotec Pfizer, New York, USA)
  Interventions: Drug: misoprostol

INTERVENTIONS:
Drug: oxytocin — 20 unit of oxytocin infusion in 500 ml lactated ringer's solution 125 ml/h (Syntocinon, Novartis, Switzerland)
  Other Names: Active Comparator
  Arms: oxytocin
Drug: misoprostol — 800 µg sublingual misoprostol (Cytotec Pfizer, New York, USA)
  Other Names: Active Comparator
  Arms: misoprostol

SUMMARY:
Researchers sought to see how oxytocin versus, sublingual misoprostol affected estimated and measured blood loss during vaginal delivery in women who had blood loss >300 ml .

DETAILED DESCRIPTION:
The greatest cause of maternal mortality globally is postpartum hemorrhage (PPH), which is defined as a blood loss of 500 mL or more after birth. All women giving birth should be given a preventive uterotonic drug, according to the World Health Organization (WHO).

Despite the use of a uterotonic drug as a preventative measure, PPH remains a frequent complication, accounting for one-quarter of all maternal fatalities worldwide. When prophylaxis fails and PPH develops, it is advised that uterotonic medicines be used as first-line therapy. However, it's unclear whether the uterotonic drug is better for treating PPH as first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* vaginal birth in women who had blood loss >300 ml

Exclusion Criteria:

* <37 weeks of pregnancy,
* genital tract injuries,
* coagulation deficit,
* hypertension, preeclampsia,
* cardiac, renal, or hepatic disease,
* epilepsy,

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — vaginal birth in women who had blood loss >300 ml
Enrollment: 150 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
measured excessive bleeding blood loss ≥ 300 mills after PPH treatment | 24 hours
  measured amount of blood loss ≥ 300 mills after PPH treatment

SECONDARY OUTCOMES:
change in hemoglobin | 12 hours
  measure change of hemoglobin
need for additional interventions | 24 hours
  number of patients need additional interventions ,like uterine aetry ligation

IPD SHARING:
Plan to Share IPD: No